CLINICAL TRIAL: NCT06420999
Title: Incidence and Impact of ICU-acquired Diaphragm Weakness
Acronym: PRODIGY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240248
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diaphragm Dysfunction
Keywords: ICU; diaphragmatic activity; Respiratory support
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients weaned from mechanical or non invasive ventilation: Adults admitted to ICU receiving either invasive mechanical ventilation for at least 48 hours, non-invasive ventilation or high-flow humidified oxygen therapy for at least 48 hours, and who have been weaned from ventilatory support within the last 24 hours.
  Interventions: Other: Diaphragmatic ultrasound and data collection

INTERVENTIONS:
Other: Diaphragmatic ultrasound and data collection — At the inclusion visit, anamnestic data available in the medical record and clinical data (vitals, chest X-ray) will be collected. At the same time, a diaphragmatic ultrasound will be performed in the half-seated position to measure diaphragmatic excursion and the thickening fraction of the right hemi-diaphragm at rest. A follow-up visit will be made on the day of discharge from intensive care, during which diaphragmatic ultrasound will be performed At D90 (+/- 15 days), the following information will be collected by consulting the electronic medical record, or by telephone if the information is not available in the record: date of discharge from hospital, date of death, date and reason for readmission to hospital or intensive care, possible introduction of long-term non-invasive ventilation, new respiratory complication after discharge from intensive care (pneumonia, atelectasis).

SUMMARY:
ICU survivors are at an increased risk of hospital and ICU readmission. Among the complications of ICU stay, diaphragmatic dysfunction is common, with a prevalence of 60 to 80%, and is associated with increased mortality and prolonged hospital stays. Furthermore, several studies have reported that the observation of impaired respiratory muscle function upon ICU discharge is associated with a poor long-term prognosis. However, the incidence and prognostic impact of persistent diaphragmatic dysfunction at ICU discharge have never been evaluated. The measurement of dyspnea, a composite evaluation of respiratory muscle function, has not been assessed for predicting prognosis upon ICU discharge.

The hypothesis of the project is that the presence of ICU-acquired diaphragmatic dysfunction at ICU discharge is associated with a poorer prognosis within 90 days.

DETAILED DESCRIPTION:
Diaphragmatic function of patients will be assessed by ultrasound within 24 hours following the weaning from ventilatory support and on the day the patient is deemed eligible for ICU discharge.

ICU discharge will be defined a priori using a checklist. Diaphragmatic activity will be assessed by bedside diaphragmatic ultrasound. Patients will be positioned in a semi-sitting position (trunk inclination between 30 and 45°) to allow for better visualization of the right hemidiaphragm. The diaphragmatic assessment will include the measurement of inspiratory and expiratory thickness to calculate the diaphragmatic thickening fraction (intercostal approach) and the measurement of diaphragmatic excursion (subcostal approach) during the respiratory cycle. These measurements will be taken at rest. Diaphragmatic dysfunction will be defined by a thickening fraction strictly less than 20% and/or a diaphragmatic excursion strictly less than 1 cm at rest.

Dyspnea will be assessed using a visual analog scale (VAS) ranging from 0 (no dyspnea) to 10 (maximum dyspnea). It will be evaluated within 24 hours following the weaning from ventilatory support and on the day the patient is deemed eligible for ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Invasive or non-invasive respiratory support (ventilation, high-flow oxygen therapy, whatever the reason) for at least 48 hours.
3. Weaning from respiratory support (invasive or not) within the last 24 hours.
4. Patient (or trusted person/relative) informed and not opposed to the study.

Exclusion Criteria:

1. Known pre-existing diaphragmatic dysfunction (phrenic lesion, neuromuscular disease, etc.)
2. Patients with tracheostomy
3. Non-communicating patients
4. Patients deprived of liberty by court or administrative order, or under legal protection (guardianship, curators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible population will be that of adult patients who have been in intensive care and have received invasive mechanical ventilation for at least 48 hours or non-invasive ventilation or humidified high-flow oxygen therapy for at least 48 hours, with a PaO2/FiO2 ratio < 200 before ventilatory support was introduced.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2028-01-29 (Estimated); Study Completion 2028-01-29 (Estimated)

PRIMARY OUTCOMES:
Association between diaphragmatic dysfunction on the day of discharge from intensive care and mortality at D90 | 90 days after inclusion (+/- 15 days)
  Mortality

SECONDARY OUTCOMES:
Association between dyspnea on the day of discharge and prognosis at D90 (composite criterion: respiratory complications, readmissions, mortality). | The day of discharge from ICU
  Measurement of dyspnea on day of discharge from intensive care, assessed by visual analog scale (VAS). Scale of 1 to 10 with 10 corresponding to minimal comfort
Quantify the proportion of patients with diaphragmatic dysfunction on the day of discharge from intensive care. | The day of discharge from ICU
  Presence of diaphragmatic dysfunction defined on ultrasound by a thickening fraction<20%.
Quantify the proportion of patients with clinically significant dyspnea on the day of discharge from intensive care. | The day of discharge from ICU
  Clinically significant dyspnea defined by a VAS>3/10. Scale of 1 to 10 with 10 corresponding to minimal comfort
Association between the presence of diaphragmatic dysfunction on the day of discharge from intensive care and length of hospital stay. | 90 days after inclusion (+/- 15 days)
  Length of hospital stay
Association between the presence of diaphragmatic dysfunction within 24 hours of weaning from ventilation and length of hospital stay. | On the day ventilation is weaned
  Presence of diaphragmatic dysfunction defined on ultrasound by a thickening fraction<20%.
Association between diaphragmatic dysfunction and the risk of hospital and intensive care readmissions | 90 days after inclusion (+/- 15 days)
  Percentage of readmissions to intensive care and hospital at D90.
Association between diaphragmatic dysfunction and the risk of respiratory complications at D90. | 90 days after inclusion (+/- 15 days)
  The percentage of respiratory complications at D90, defined by the occurrence of pneumonia, reintubation, atelectasis (or worsening in case of pre-existing abnormality).

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine intensive Réanimation, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.